CLINICAL TRIAL: NCT03926624
Title: Phase 3 Randomized Trial of DFP-10917 vs Non-Intensive Reinduction (LoDAC, Azacitidine, Decitabine, Venetoclax Combination Regimens) or Intensive Reinduction (High & Intermediate Dose Cytarabine Regimens) for Acute Myelogenous Leukemia Patients in Second, Third, or Fourth Salvage
Brief Title: Trial of DFP-10917 vs Non-Intensive or Intensive Reinduction for AML Patients in 2nd/3rd/4th Salvage
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The data met the protocol-specified criteria for futility of the investigational treatment.
Sponsor: Delta-Fly Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D18-11141
Record Dates: First submitted 2019-04-11; First posted 2019-04-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-02

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — DFP-10917; Cytarabine; Azacitidine; Decitabine; Mitoxantrone; Etoposide; fludarabine; Idarubicin; venetoclax; Cladribine

STUDY DESIGN:
Intervention Model Description: randomized, controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): DFP-10917 Dose: 6 mg/m²/day administered by continuous infusion for 14 days followed by a 14-day resting period per 28-day treatment cycle. If a patient experiences a significant treatment-related AE, the patient may undergo one dose reduction of DFP-10917 to 4 mg/m²/day x 14 days for subsequent treatment cycles
  Interventions: Drug: DFP-10917
- Control (Active Comparator): Non-Intensive:
  * LoDAC: 20 mg SC BID 10 days
  * Azacitidine: 75 mg/m²/day SC 7 days(or 5+2)
  * Decitabine: CIV 20 mg/m²x5 days
  * Venetoclax + LoDAC/Azacitidine/Decitabine:LoDAC-Venetoclax ramp-up to 600 mgxday. Cytarabine SC 20 mg/m²xday D1-10. Azacitidine or Decitabine-Venetoclax ramp-up to 400 mgxday. Azacitidine IV or SC 75 mg/m² D1-7. Decitabine IV 20 mg/m² on D1-5 or 1-10.
  Intensive:
  * High DAC: cytarabine 1-2 g/m² up to 5 days, max total dose 10 g/m²
  * FLAG: D1-5: fludarabine 30 mg/m² IV for 30min, D1-5: cytarabine 1-2 g/m² for 4hr daily x 5 & G-CSF 5 mcg/kg or 300 mcg/m² until PMN recovery, with or without idarubicin D1-3 8 mg/m² IV dailyx3 (FLAG-Ida)
  * MEC: D1-6: mitoxantrone 6 mg/m² IV bolus, etoposide 80 mg/m² IV 1hr & cytarabine 1g/m² IV 6hr.
  * CLAG/M or Ida = cladribine 5 mg/m² D1-5, cytarabine 2 g/m² D1-5, G-CSF 300 μg D0-5, mitoxantrone 10 mg/m² D1-3 or Idarubicin 10 mg/m² D1-3.
  * Intermediate DAC: cytarabine 20 mg/m² IV dailyx5
  Interventions: Drug: Cytarabine; Drug: Azacitidine; Drug: Decitabine; Drug: Mitoxantrone; Drug: Etoposide; Drug: Fludarabine; Drug: Idarubicin; Drug: Venetoclax; Drug: Cladribine

INTERVENTIONS:
Drug: DFP-10917 — DFP-10917 Powder for Injection. Active ingredient: 4-amino-1-(2-cyano-deoxy-β-D-arabinofuranosyl)-2(1H)-pyrimidinone monohydrochloride
  Arms: Experimental
Drug: Cytarabine — cytosine arabinoside (ara-C)
  Arms: Control
Drug: Azacitidine — Azacitidine
  Arms: Control
Drug: Decitabine — Decitabine
  Arms: Control
Drug: Mitoxantrone — Mitoxantrone
  Arms: Control
Drug: Etoposide — Etoposide
  Arms: Control
Drug: Fludarabine — Fludarabine
  Arms: Control
Drug: Idarubicin — Idarubicin
  Arms: Control
Drug: Venetoclax — Venetoclax
  Arms: Control
Drug: Cladribine — Cladribine
  Arms: Control

SUMMARY:
Phase III, multicenter, randomized study with two arms (1:1 ratio) enrolling patients with AML relapsed/refractory after 2, 3, or 4 prior induction regimens:

Experimental arm: DFP-10917 14-day continuous intravenous (IV) infusion at a dose of 6 mg/m²/day followed by a 14-day resting period per 28-day cycles.

Control arm: Non-Intensive Reinduction (LoDAC, Azacitidine, Decitabine, Venetoclax Combination Regimens) or Intensive Reinduction (High and Intermediate Dose Cytarabine Regimens), depending on the patient's prior induction treatment.

DETAILED DESCRIPTION:
Study to compare the rate of complete response (CR) and duration of CR, in patients with relapsed or refractory AML to two, three, or four prior induction regimens that may have included intensive chemotherapy (e.g., "7+3" cytarabine and daunorubicin), epigenetic therapy (i.e., azacitidine or decitabine), or targeted therapy (e.g., FLT-3, IDH-1/2, BCL-2, monoclonal antibody), who will receive DFP-10917 versus non-intensive reinduction (LoDAC, azacitidine, decitabine, venetoclax + LoDAC or azacitidine or decitabine) or intensive reinduction (high and intermediate dose cytarabine regimens) as a second, third, or fourth salvage treatment.

Experimental Arm DFP-10917 Dose: 6 mg/m²/day administered by continuous infusion for 14 days followed by a 14-day resting period per 28-day treatment cycle. If a patient experiences a significant treatment-related AE, the patient may undergo one dose reduction of DFP-10917 to 4 mg/m²/day x 14 days for subsequent treatment cycles

Control arm: Non-Intensive Reinduction (LoDAC, Azacitidine, Decitabine, Venetoclax + LoDAC or Azacitidine or Decitabine) or Intensive Reinduction (High and Intermediate Dose Cytarabine Regimens), depending on the patient's prior induction treatment as well as the patient's clinical condition and comorbidities. Control treatment is to be selected only from among the following. Institutional practice for administering these treatments are permitted, but the dose and days of drug administration should be followed as below.

Non-Intensive Reinduction:

* LoDAC: 20 mg Cytarabine administered by subcutaneous (SC) injection, twice daily (BID) for 10 days, plus best supportive care per 28-day treatment cycle
* Azacitidine: 75 mg/m²/day administered by SC for 7 consecutive days (or 5+2), plus best supportive care per 28-day treatment cycle
* Decitabine: administered as continuous intravenous (CIV) infusion 20 mg/m² x 5 days plus best supportive care per 28 day treatment cycle
* Venetoclax + LoDAC or Azacitidine or Decitabine: In combination with LoDAC, Venetoclax will be administered via a daily ramp-up to a final 600 mg once daily dose. During the ramp-up, patients are to receive TLS prophylaxis and may be hospitalized for monitoring. Cytarabine will be administered subcutaneously at a dose of 20 mg/m² once daily on Days 1-10 of each 28-day cycle beginning Cycle 1 Day 1. In combination with Azacitidine or Decitabine, Venetoclax will be administered via a daily ramp-up to a final 400 mg once daily dose. Azacitidine will be administered intravenously or subcutaneously at a dose of 75 mg/m² on Days 1-7 of each 28-day cycle beginning on Cycle 1 Day 1. Decitabine will be administered via IV at a dose of 20 mg/m² on Days 1-5 or 1-10, as per institutional practice, of each 28-day cycle beginning Cycle 1 Day 1.

Intensive Reinduction:

* High DAC = cytarabine at doses of 1-2 g/m²/day for up to 5 days, with a maximum total dose 10 g/m² per course
* FLAG = Days 1-5: fludarabine 30 mg/m² IV over 30 minutes, Days 1-5: cytarabine 1 2 grm/m² over 4 hours daily x 5, and granulocyte colony-stimulating factor 5 mcg/kg or 300 mcg/m² until Polymorphonuclear Neutrophil (PMN) recovery, with or without idarubicin Days 1-3 at 8 mg/m² IV daily x 3 (FLAG-Ida)
* MEC = Days 1-6: mitoxantrone 6 mg/m² IV bolus, etoposide 80 mg/m² IV over 1 hour, and cytarabine 1 grm/m² IV over 6 hrs (Etoposide may be deleted per institutional guidelines, i.e., HAM regimen)
* CLAG/M or Ida = cladribine 5 mg/m² on Days 1-5, cytarabine 2 g/m² on Days 1-5, granulocyte-colony stimulating factor 300 μg on Days 0-5 (G-CSF starts 24 hr prior to chemotherapy), and mitoxantrone 10 mg/m² on Days 1-3 or Idarubicin 10 mg/m² on Days 1-3
* Intermediate DAC = cytarabine 20 mg/m² IV daily x 5

The selection of control arm treatment will be determined by the investigator depending on the patient's prior initial induction and salvage treatment regimen(s), as well as the patient's clinical condition and comorbidities. The investigator will select the patient's control treatment from among the non-intensive or intensive regimens prior to study treatment randomization in order to balance treatment allocation between the experimental and control treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or pathologically confirmed diagnosis of AML based on WHO classification that has relapsed after, or is refractory to, two, three, or four prior induction regimens that may have included intensive chemotherapy (e.g., "7+3" cytarabine and daunorubicin), epigenetic therapy (i.e., azacitidine or decitabine), or targeted therapy (e.g., FLT-3, IDH-1/2, BCL-2, monoclonal antibody).

   (Relapse is defined as reemergence of ≥5% leukemia blasts in bone marrow or ≥1% blasts in peripheral blood ≥90 days after first CR or CR without complete platelet recovery (CRp). Refractory AML is defined as persistent disease ≥28 days after initiation of intensive induction therapy (up to two induction cycles) or relapse <90 days after first CR or CRp. Refractory disease for patients undergoing hypomethylating agent induction is defined as lack of remission following at least 2 cycles of epigenetic therapy without reduction in bone marrow blast status.)

   Patients with a history of IPSS-R high or very high risk MDS that transformed to AML during treatment with hypomethylating drugs and then relapse following or are refractory to a subsequent AML induction regimen may be enrolled as Second Salvage AML patients. Additionally, patients with a history of MPN in accelerated phase (MPN-AP) or high-risk primary myelofibrosis (PMF) that transformed to AML during treatment with hypomethylating drugs and then relapse following or are refractory to a subsequent AML induction regimen may be enrolled as Second Salvage AML patients.
2. Aged ≥ 18 years.
3. ECOG Performance Status of 0, 1 or 2.
4. Adequate clinical laboratory values (i.e., plasma creatinine <2.5 x upper limit of normal (ULN) for the institution, bilirubin <2.5 x ULN, alanine transaminase (ALT) and aspartate transaminase (AST) ≤2.5 x ULN).
5. Absence of active central nervous system (CNS) involvement by leukemia. Patients with previously diagnosed CNS leukemia are eligible if the CNS leukemia is under control and intrathecal treatment may continue throughout the study.
6. Absence of uncontrolled intercurrent illnesses, including uncontrolled infections, cardiac conditions, or other organ dysfunctions.
7. Signed informed consent prior to the start of any study specific procedures.
8. Women of child-bearing potential must have a negative serum or urine pregnancy test.
9. Male and female patients must agree to use acceptable contraceptive methods for the duration of the study and for at least one month after the last drug administration.

Exclusion Criteria:

1. The interval from prior treatment to time of study drug administration is < 2 weeks for cytotoxic agents or < 5 half-lives for noncytotoxic agents. Exceptions: Use of hydroxyurea is allowed before the start of study and is to be discontinued prior to the initiation of study treatment. At the investigator's discretion, for patients with significant leukocytosis that develops during the early treatment cycles, hydroxyurea may be administered. The hydroxyurea should be discontinued as soon as clinically appropriate.
2. Any >grade 1 persistent clinically significant toxicities from prior chemotherapy.
3. Inadequate Cardiac (left ventricular ejection fraction ≤40%) function.
4. White blood cell (WBC) count >15,000/μL (Note: Patients considered for possible venetoclax-containing regimen must have WBC ≤10k/μL prior to initiating venetoclax treatment).
5. For patients with prior hematopoietic stem cell transplant (HSCT):

   1. Less than 3 months since HSCT
   2. Acute Graft versus Host Disease (GvHD) >Grade 1
   3. Chronic GvHD >Grade 1
6. Any concomitant condition that in the opinion of the investigator could compromise the objectives of this study and the patient's compliance.
7. A pregnant or lactating woman.
8. Current malignancies of another type. Exceptions: Patients may participate if they have previously treated and currently controlled prostate cancer, or adequately treated in situ cervical cancer or basal cell skin cancer, or other malignancies with no evidence of disease for 2 years or more.
9. Patient has acute promyelocytic leukemia (APL).
10. Patients with known HIV, active HBV or active HCV infection (note: testing for these infections is not required). For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
11. Documented or known clinically significant bleeding disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
Complete remission (CR) rate | 3 years
  The rate of CR based on International Working Group (IWG) Guidelines for bone marrow and blood response
Duration of complete remission | 3 years
  Number of days from time of initial CR until disease recurrence or death

SECONDARY OUTCOMES:
The rate of complete remission (CR) + (complete remission with incomplete hematologic recovery) CRi+ (complete remission with partial hematologic recovery) CRp | 3 years
  CR as above including neutrophil granulocyte count > 0.5x10^9/L & platelet count > 50x10^9/L
The duration of complete remission (CR) + (complete remission with incomplete hematologic recovery) CRi+ (complete remission with partial hematologic recovery) CRp | 3 years
  CR as above including neutrophil granulocyte count > 0.5x10^9/L & platelet count > 50x10^9/L + platelet count < 100x10^9/L
Overall survival | 3 years
  Number of days from date of first dose to date of death
Transition rate to hematopoietic stem cell transplantation (HSCT) | 3 years
  Number of subjects who transition to HSCT
Overall response rate (ORR) | 3 years
  The rate of CR + CRi + CRp + PR
Duration overall response | 3 years
  The duration of CR + CRi + CRp + PR
Rate of disease related co-morbidities | 3 years
  Number and severity of expected leukemia-related adverse events
Adverse events | 3 years
  Number of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tapan Kadia, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (39):
- United States (39):
  - O'Neal Comprehensive Cancer Center, Birmingham, Alabama
  - Banner MD Anderson, Gilbert, Arizona
  - HonorHealth (VGPCC Cancer Transplant Institute), Scottsdale, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - University of California, Irvine, California
  - UCLA, Los Angeles, California
  - UF-Health Cancer Center Gainesville, Gainesville, Florida
  - Baptist MD Anderson, Jacksonville, Florida
  - UF-Health Jacksonville, Jacksonville, Florida
  - AdventHealth Medical Group Blood and Marrow Transplant at Orlando, Orlando, Florida
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Rush University, Chicago, Illinois
  - Decatur Memorial Hospital-Cancer Care Specialists of Central IL, Decatur, Illinois
  - Loyola University Medical Center, Hines, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - The University of Kansas Cancer Center, Westwood, Kansas
  - University of KY- Markey Cancer Center, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Ochsner Benson Cancer Center, Jefferson, Louisiana
  - Tulane University, New Orleans, Louisiana
  - Henry Ford Cancer Institute, Detroit, Michigan
  - The University of Mississippi Medical Center, Jackson, Mississippi
  - New York Medical College, Valhalla, New York
  - Novant Health Cancer Institute - Elizabeth (Hematology), Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Vidant Oncology, Kinston, North Carolina
  - Novant Health Cancer Institute - Forsyth (Hematology), Winston-Salem, North Carolina
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - Seidman Cancer Center, University Hospitals, Cleveland Medical Center, Cleveland, Ohio
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Avera Medical Group, Sioux Falls, South Dakota
  - UT Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - Multicare Institute for Research and Innovation, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No